CLINICAL TRIAL: NCT03890406
Title: The Effect of Deep Neuromuscular Blockade on Requirement of Intravenous Anesthetic Agent During Laparoscopic Colorectal Surgery
Brief Title: The Effect of Deep Neuromuscular Blockade on Requirement of Intravenous Anesthetic Agent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, BON WOOK KOO, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEEPTIVA
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Laparoscopy; General Anesthesia; Neuromuscular Blockade
Keywords: Deep neuromuscular blockade

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Experimental): Deep neuromuscular blockade
  Interventions: Drug: Rocuronium: PTC(Post-tetanic count) 1~2
- Group M (Active Comparator): Moderate neuromuscular blockade
  Interventions: Drug: Rocuronium: TOF(Train-of-four) 1~2

INTERVENTIONS:
Drug: Rocuronium: PTC(Post-tetanic count) 1~2 — Deep neuromuscular blockade will be maintained using continuous infusion of rocuronium.
  Other Names: Deep block
  Arms: Group D
Drug: Rocuronium: TOF(Train-of-four) 1~2 — Moderate neuromuscular blockade will be maintained using continuous infusion of rocuronium.
  Other Names: Moderate block
  Arms: Group M

SUMMARY:
Recently, deep neuromuscular blockade during general anesthesia has been studied by many authors regarding various effects upon patients' outcomes and surgical conditions. We believe deep neuromuscular blockade can be especially beneficial in laparoscopic surgery, because it can expand surgical space and prevent patients' minute movements that can disturb precise operations. In clinical situations, anesthetists tend to compensate the insufficiency of neuromuscular blockade by increasing the dose of other anesthetic agents, which can prolong patients' recovery time and impair the surgical condition. In this study, we plan to divide the patients into 2 groups according to the depth of neuromuscular blockade, and compare the dose of anesthetic agent used to maintain surgical condition.

DETAILED DESCRIPTION:
Patients undergoing elective laparoscopic colorectal surgery are going to be recruited and divided into 2 groups: Group D will receive deep neuromuscular blockade, and Group M will receive moderate neuromuscular blockade using continuous infusion of rocuronium. Acceleromyography(TOF-watch SX) will be used to monitor the depth of blockade. In both groups, the anesthesia will be maintained with TIVA(total intra-venous anesthesia) including continuous target-controlled infusion of propofol and remifentanil. During the surgery, the number of patient movement and restoration of self respiration will be recorded. At the end of anesthesia, the dose of propofol and remifentanil used will be assessed and compared between the groups. Also, the satisfaction score of surgeons regarding the surgical condition, the anesthesia time, the operation time will be documented. After the patients are discharged, their charts are going to be reviewed and whether any pulmonary or surgical complications occurred will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic colorectal resection due to benign or malignant neoplasm of colon or rectum
* ASA class I or II

Exclusion Criteria:

* Patients receiving medications known to have drug-drug interaction with neuromuscular blocking agents
* Patients who have significantly impaired cardiac, pulmonary, hepatic, renal function
* Patients who are pregnant
* Patients who are known to have hypersensitivity to the anesthetic/analgesic/neuromuscular blocking agents which are going to be used in the study
* BMI < 18.5 or > 35.0 kg/m2
* Patients with previous history of open abdominal surgery
* Patients with previous history of malignant hyperthermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Dosage of propofol | intraoperative (from starting of anesthesia to end of anesthesia)
  the amount of propofol used (mg/kg)

SECONDARY OUTCOMES:
Dosage of remifentanil | intraoperative (from starting of anesthesia to end of anesthesia)
  the amount of remifentanil used (mcg/kg)
Patient movement | intraoperative (from tracheal intubation to injection of neuromuscular reversal agent)
  the observed number of patient movement during the surgery
Patient self respiration | intraoperative (from tracheal intubation to injection of neuromuscular reversal agent)
  the observed number of restoration of self breathing during the surgery (ex. EtCO2 notching)
Surgical condition score | assessed at the end of the surgery
  the 5-point satisfaction score of surgeon regarding surgical conditions

CONTACTS AND LOCATIONS:
Overall Officials: Ah Young Oh, MD, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Nam SW, Oh AY, Koo BW, Kim BY, Han J, Chung SH. Effects of depth of neuromuscular blockade on the BIS-guided propofol requirement: A randomized controlled trial. Medicine (Baltimore). 2021 Jul 23;100(29):e26576. doi: 10.1097/MD.0000000000026576. PMID 34398011